CLINICAL TRIAL: NCT00530192
Title: A Pilot Study Utilizing Molecular Profiling of Patients' Tumors to Find Potential Targets and Select Treatments for Their Refractory Cancers
Brief Title: Molecular Profiling Protocol (SCRI-CA-001)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Scottsdale Healthcare (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Scottsdale Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI-CA-001; SCRI-CA-001
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Refractory Cancer
Keywords: Refractory Cancer; Molecular Profile
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Treatment based on Molecular Profiling — Treatment with commercially available treatments (per package insert instructions)

SUMMARY:
This is an open-label, multicenter pilot study in patients with advanced solid tumors.

The primary objective of this study is to compare progression-free survival using a treatment regimen selected by molecular profiling with progression-free survival for the most recent regimen the patient has progressed on.

To be eligible, patients must have received at least two lines of prior chemotherapeutic, hormonal or biological regimens for advanced disease, have measurable or evaluable, refractory disease and have clear documentation of the time between treatment start and documented progression on the last treatment prior to study entry. Eligible patients must undergo or have available a tumor biopsy for molecular profiling within 2 months of IHC/FISH and/or DNA microarray analysis.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer which has progressed on 2 prior chemotherapeutic, hormonal or biological regimens for advanced disease.
* Be defined as refractory to the last line of therapy
* Have documentation of the best clinical response to the treatment regimen immediately prior to entering this study

Exclusion Criteria:

* Patients with symptomatic CNS metastasis
* Any previous history of another malignancy within 5 years of study entry
* Uncontrolled intercurrent illness
* Known HIV, HBV, HCV infection
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03

PRIMARY OUTCOMES:
To compare progression-free survival using a treatment regimen selected by molecular profiling with progression-free survival for the most recent regimen the patient has progressed on. | Every 8 weeks disease assessments are performed

SECONDARY OUTCOMES:
To determine the frequency with which molecular profiling of a patient's tumor by IHC/FISH and/or microarray analysis yields a target against which there is a commercially available, approved therapeutic regimen. | Time of Profiling- Baseline
To determine the response rate (according to RECIST or disease-specific response criteria) and the percent of patients with non-progression at 4 months in patients with solid tumors whose therapy is selected by molecular profiling. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Von Hoff, MD, Principal Investigator — TGen Clinical Research Services at Scottsdale Healthcare
Locations (9):
- United States (9):
  - Oncology Specialties, Huntsville, Alabama
  - TGen Clinical Research Services, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Tower Oncology, Beverly Hills, California
  - Louis Warschaw Prostate Cancer Center at Cedars Sinai Medical Center, Los Angeles, California
  - Central Indiana Cancer Center, Indianapolis, Indiana
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - South Texas Oncology Hematology, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas